CLINICAL TRIAL: NCT05993897
Title: Effect of Sodium Glucose Co-transporter 2 Inhibitors on Left Atrium Remodeling in Non-valvular Paroxysmal Atrial Fibrillation Patients
Brief Title: Effect of Sodium Glucose Co-transporter 2 Inhibitors on Left Atrial Remodeling
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Aswan University (Other)
Responsible Party: Principal Investigator, Aml Soliman, Lecturer of cardiology, Aswan university, Aswan University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 693/11/22
Record Dates: First submitted 2023-07-25; First posted 2023-08-15 (Actual); Last update posted 2023-08-15 (Actual); Status verified 2023-08

CONDITIONS: Atrial Fibrillation
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Dapagliflozin (Active Comparator): patients who will receive SGLT2 inhibitors
  Interventions: Drug: Sodium Glucose Co-transporter 2 (SGLT2) Inhibitor; Drug: Rhythm control and anticoagulation
- Placebo (Placebo Comparator): Patients who will receive Rhythm control +/- oral anticoagulation
  Interventions: Drug: Rhythm control and anticoagulation

INTERVENTIONS:
Drug: Sodium Glucose Co-transporter 2 (SGLT2) Inhibitor — 10 mg of Dapagliflozin orally once daily
  Arms: Dapagliflozin
Drug: Rhythm control and anticoagulation — In acute stage: Cardioversion with D.C shock if haemodynamically unstable, after failure of pharmacological cardioversion or participant preference.
  or pharmacological cardioversion with either IV cordarone in structurally abnormal heart (150mg over 10 minutes followed by1 mg/min infusion for 6 hours followed by 0.5 mg/min not exceeding 2.4 grams over 24 hours till restoration of sinus Rhythm. Then maintenance dose of 200 mg tab orally every 8 hours for 3 weeks then 200 mg tab orally once per day.
  or Propafenone (Rytmonorm) 600 mg single oral dose in structurally normal heart then maintenance dose of 150mg tab orally every 8 hours.
  + Rivaroxaban 20mg orally once daily if CHA2DS2 VASc score 1 or more for males and 2 or more for females.

SUMMARY:
Investigators are going to assess direct effect of SGLT2 inhibitors on left atrial remodeling in participants with nonvalvular paroxysmal atrial fibrillation regardless of diabetes status.

ELIGIBILITY:
Inclusion Criteria:

1. with non-valvular paroxysmal atrial fibrillation (AF that terminates spontaneously or with intervention within seven days of onset).
2. Patient age 18-60 years.
3. Patients with Glomerular Filtration Rate (GFR) >45 ml/min/1.73m2 (Cockcroft-Gault equation).
4. Patient with normal left atrium or dilated (diameter <5 cm)

Exclusion Criteria:

1. Patients < 18 yrs old.
2. Patients with valvular heart diseases (Moderate to severe MS, severe AS, Prosthetic heart valves).
3. Patients with left atrium > 5cm.
4. Patients with glomerular Filtration Rate (GFR) <45 ml/min/1.73m2 (Cockcroft-Gault equation).
5. Patient with ischemic heart disease (previous MI, UA, PCI or CABG).
6. Patient with previous ischemic stroke.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2023-08 (Estimated); Primary Completion 2024-08 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Left atrial remodeling | Before first administration of treatment and will be repeated 6 months after while still on treatment
  by measuring Indexed LA volume (LAVI) in ml/m2
Changes in left atrial strain | Before first administration of treatment and will be repeated 6 months after while still on treatment
  by measuring left atrial strain %
Changes in left atrial systolic force | Before first administration of treatment and will be repeated 6 months after while still on treatment
  by measuring left atrial systolic force in ml/m3

SECONDARY OUTCOMES:
Mean percentage of time spent in atrial fibrillation | After the first dose of treatment till the end of the study (1 year)
  By documented ECG or Holter monitoring
Mortality Rate | After the first dose of treatment till the end of the study (1 year)
  all cause mortality
Incidence of Hospitalization due to HF | After the first dose of treatment till the end of the study (1 year)
  In hospital admission by HF symptoms
Number of participants with Stroke | After the first dose of treatment till the end of the study (1 year)
  Ischemic or hemorrhagic

IPD SHARING:
Plan to Share IPD: No